CLINICAL TRIAL: NCT01620684
Title: The Effects of Cortisol Blockade on Nutritional Sympathetic Nervous System Responsiveness in Overweight and Obese Subjects With Metabolic Syndrome
Brief Title: Cortisol and Nutritional Sympathetic Responsiveness
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Baker Heart Research Institute (Other)
Responsible Party: Principal Investigator, Nora E. Straznicky, Senior Research Officer, Baker Heart Research Institute
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Metyrapone; Heart Foundation G11M5892 (Other Grant/Funding Number: Heart Foundation of Australia)
Record Dates: First submitted 2012-06-12; First posted 2012-06-15 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Metabolic Syndrome; Obesity; Insulin Resistance
MeSH Terms: conditions — Metabolic Syndrome; Obesity; Insulin Resistance | interventions — Metyrapone; lactitol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- metyrapone (Active Comparator): Overnight metyrapone treatment (total dose of 30 mg/kg)
  Interventions: Drug: metyrapone
- sugar pill (Placebo Comparator): Overnight treatment with placebo capsules
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: metyrapone — Overnight treatment (15 mg/kg at midnight and 15 mg/kg at 6 am)
  Other Names: Metopirone (Novartis)
  Arms: metyrapone
Drug: placebo — placebo capsules
  Arms: sugar pill

SUMMARY:
This project will examine whether short-term (over a 12-hour period) pharmacological lowering of the stress hormone 'cortisol' improves the nervous system response to food intake in overweight or obese individuals who have metabolic syndrome.

The investigators know from our previous research that overweight/obese persons who are insulin resistant, have a blunted sympathetic nervous response to carbohydrate ingestion. This means that they are less able to dissipate energy from caloric intake, which would favour the maintenance of the obese state. Cortisol adversely impacts on insulin action and transport into the brain and cortisol levels are often elevated in persons with central (abdominal) obesity.

A randomized, double-blind, placebo controlled, cross-over design will be used to compare the effects of overnight treatment with metyrapone (15 mg/kg at midnight and 15 mg/kg at 6 am) versus placebo on sympathetic nervous system activity in response to a standard 75-g oral sugar (glucose) tolerance test. A 2 week washout will separate treatments.

Metyrapone is a drug that reversibly inhibits the enzyme 11beta-hydroxylase, and therefore the production of cortisol. It is used clinically to test the activity of the adrenal gland (the key site of cortisol production) and the pituitary gland. The investigators anticipate that at the dosage used, it will lower blood cortisol concentration by 44 to 64% during the experimental morning.

The study protocol comprises two screening visits and two experimental mornings. Key procedures will include:

* Assessment of insulin action (sensitivity) using the gold standard 'clamp' method.
* Measurement of sympathetic nervous system activity by both biochemical methods (isotope dilution which provides a measure of the apparent rate of release of 'noradrenaline'-the key neurotransmitter in the sympathetic nervous system) and direct intra-neuronal nerve recordings from the peroneal nerve in the lower leg.
* Indirect calorimetry to assess resting metabolic rate and the response to sugar ingestion.
* DEXA scan to quantify fat and lean mass.
* Assessment of arterial elasticity and calf blood flow by non-invasive methods.
* A standard 75g oral sugar tolerance test.

The results will provide important new information regarding the role of cortisol on nervous system function in overweight/obese individuals.

DETAILED DESCRIPTION:
Similarities between metabolic syndrome obesity and hypercortisolemic conditions such as Cushing's syndrome have raised interest in the pathogenic role of glucocorticoid excess in this clinical setting. Cortisol is a well known counter-regulator of insulin action and increased levels of serum cortisol have been linked to insulin resistance in many studies. Moreover, treatment with the synthetic glucocorticoid dexamethasone reduced central nervous system insulin uptake by 49% in dogs. We have previously identified in metabolic syndrome subjects, an inverse relationship between morning fasting cortisol levels and sympathetic neural responsiveness to oral glucose ingestion. This concurs with other evidence that cortisol and synthetic glucocorticoids have sympathoinhibitory effects.

This project will test the hypothesis that short-term lowering of plasma cortisol levels by overnight metyrapone treatment, will improve nutritional sympathetic nervous system responses to carbohydrate ingestion in obese insulin resistant subjects with metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* un-medicated,
* overweight or obese subjects (12 men and 12 postmenopausal women),
* weight-stable,
* non-smoking,
* aged 45-65 years
* will be recruited on the basis of having > 3 MetS criteria as per the newly harmonized definition.
* elevated waist circumference will be defined as > 102 cm in men and > 88 cm in women.
* all subjects will also be insulin resistant (HOMA index > 2.5 and/or euglycaemic hyperinsulinemic clamp derived M/I value < 8 mg per kg fat free mass per minute per mU/L x 100).

Exclusion Criteria:

* adrenocortical insufficiency,
* pituitary dysfunction or tumour,
* sleep apnoea treated with CPAP,
* cardiovascular disease (previous MI, angina, stroke, heart failure, secondary hypertension),
* renal or hepatic disease (serum creatinine > 0.2 mmol/L; > 1 proteinuria on dipstick; alanine transferase > 2.5 times upper limit of normal, active liver disease) or
* diseases which may affect measured parameters (e.g. thyroid, Cushing's or Addison's diseases).

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Nutritional sympathetic nervous system responsiveness | 12-hours
  Effects of acute overnight metyrapone treatment will be studied

SECONDARY OUTCOMES:
insulin sensitivity | 12 hours
  Acute effects of overnight metyrapone treatment will be studied

CONTACTS AND LOCATIONS:
Overall Officials: Nora E Straznicky, PhD MPH, Principal Investigator — Baker IDI Heart & Diabetes Institute
Locations (1):
- Heart Centre, Alfred Hospital, Prahran, Melbourne, Victoria, Australia